CLINICAL TRIAL: NCT07291921
Title: Development of a Non-Invasive Postoperative Recurrence Monitoring Method for Lung Cancer After Neoadjuvant Immunotherapy
Brief Title: Non-Invasive Postoperative Recurrence Monitoring After Neoadjuvant Immunotherapy in Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Chen KeZhong, Professor, Peking University People's Hospital
Other Study IDs: BRWEP2024W034080204-1
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Lung Neoplasms; Neoadjuvant Therapy; Immunotherapy; Minimal Residual Disease
Keywords: NSCLC; Neoadjuvant immunotherapy; Perioperative monitoring; Liquid biopsy; MRD; Minimal residual disease; Multiple omics
MeSH Terms: conditions — Lung Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-risk group: High-risk recurrence groups identified by the multi-omics model
- Low-risk group: Low-risk recurrence groups identified by the multi-omics model

SUMMARY:
This project aims to innovatively integrate multi-omics data, including plasma metabolomics, radiomics, and cfDNA multi-level information, combined with survival data (e.g., RFS), to establish a novel multidimensional approach for noninvasive postoperative recurrence monitoring in lung cancer using artificial intelligence algorithms. The goal is to develop a new noninvasive recurrence monitoring system for lung cancer.

DETAILED DESCRIPTION:
This project is a prospective observational study designed to comprehensively integrate plasma metabolomic, radiomic, and epigenomic data to develop a predictive model for postoperative recurrence risk in lung cancer. The study will retrospectively enroll 200 patients who underwent radical surgery after neoadjuvant therapy, and prospectively enroll 100 additional post-radical-surgery lung cancer patients who received neoadjuvant treatment as a validation cohort. Peripheral blood samples will be collected at multiple timepoints for metabolomic profiling. Unsupervised clustering, random forest algorithms, and Wilcoxon tests will be applied to identify recurrence-related features and construct a recurrence prediction model.Additionally, using preoperative and first postoperative follow-up CT imaging data, a deep learning-based 3D ResNet will be employed to generate radiomic recurrence risk scores for each patient. Plasma cfDNA will undergo low-pass whole-genome sequencing and methylation analysis to extract multi-dimensional recurrence-associated features. Finally, the study will innovatively utilize the DeepProg deep learning framework to integrate radiomic, cfDNA, and plasma metabolomic data into a non-invasive multi-omics model. Combined with survival data, this model will predict recurrence risk, ultimately achieving high-accuracy stratification of patients' postoperative recurrence probability.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Male or female, aged ≥ 18 and < 85 years.
3. Radical resection performed, pathologic stage IB-IIIA (8th TNM) non-small-cell lung cancer.
4. Tumor tissue and blood samples obtainable at all protocol-specified time-points.
5. No pure ground-glass nodule on imaging.
6. Completed standard neoadjuvant immunotherapy combined with platinum-based chemotherapy.

Exclusion Criteria:

1. Postoperative pathology shows other than NSCLC, including but not limited to benign lesions, small-cell carcinoma, metastasis, or indeterminate/inadequate histology.
2. Insufficient or poor-quality blood or tissue samples.
3. Pure ground-glass nodule on imaging.
4. History of any malignancy within the past 5 years.
5. Contraindication to surgery preventing radical resection.
6. Non-radical (R2) resection.
7. Pathologic stage IIIB-N3, IIIC, or IV on paraffin sections.
8. Refusal or withdrawal of informed consent.
9. Any condition deemed unsuitable by the investigator (e.g., perioperative blood transfusion, severe psychiatric disorder precluding follow-up).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary nodules who underwent radical treatment at our center between May 2025 and October 2027, met all eligibility criteria, and provided informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Two-year recurrence-free survival rate | Time from curative surgery to confirmation of clinical progression (recurrence or metastasis) within two years

SECONDARY OUTCOMES:
Overall survival | Time from curative surgery to confirmation of death (any cause)，assessed up to 60 months.
Timely diagnosis rate by the novel MRD monitoring technique | two years
  The proportion of patients with recurrence signals detected by non-invasive methods prior to clinical confirmation of recurrence/metastasis, and quantify the mean lead time.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided